CLINICAL TRIAL: NCT06595680
Title: Development of an Innovative Hemodialysis Method to Improve Dialytic Clearance of Protein-bound Uremic Toxins
Acronym: CLEARTOX
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL23_0031; 2023-510406-41-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: End Stage Renal Disease; Chronic Hemolysis
Keywords: End stage renal disease; Hemodialysis; Protein Bound Uremic Toxins; p-Cresyl Sulfate; Indoxyl Sulfate; Medium Chain fatty acids; Medium chain triglycerides; Octanoate; Decanoate; Medialipide
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Perfusion; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Each patient will sequentially receive during two 4 hours hemodialysis session separated by one week a perfusion of Medialipide and a perfusion of NaCl 0,9%. The order of intervention will be determined by randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medialipide 20% - NaCl 0,9% (Experimental): Group 1 will receive during the first interventional hemodialysis session a perfusion of Medialipide 20% perfused at a rate of 0,11 gram/kilogram/hour (g/kg/h) during 4 hours. One week late, they will receive during the second interventional hemodialysis session a perfusion of NaCl 0,9% with a volume corresponding to the one of Medialipide also during 4 hours.
  Interventions: Drug: Medialipide 20% perfusion; Drug: NaCl 0,9%; Biological: Blood sample
- NaCl 0,9% - Medialipide 20% (Experimental): Group 2 will receive during the first interventional hemodialysis session a perfusion of NaCl 0,9% with a volume corresponding to the one of Medialipide during 4 hours. One week late, they will receive during the second interventional hemodialysis session a perfusion of Medialipide 20% perfused at a rate of 0,11 gram/kilogram/hour (g/kg/h) also during 4 hours.
  Interventions: Drug: Medialipide 20% perfusion; Drug: NaCl 0,9%; Biological: Blood sample

INTERVENTIONS:
Drug: Medialipide 20% perfusion — Each patient will receive during a 4 hours hemodialysis session a perfusion of Medialipide 20% at a rate of 0,11 g/kg/h. Medialipide will be perfused using the venous line connected to the hemodialysis machine.
Drug: NaCl 0,9% — Each patient will receive during a 4 hours hemodialysis session a perfusion of NACL 0,9% with a volume corresponding to the one of Medialipide 20%. NaCl 0,9% will be perfused using the venous line connected to the hemodialysis machine.
Biological: Blood sample — Serial biological sampling for the measurement of different blood concentrations : electrolytes, serum protein , albumin, renal function (urea, creatinine), hemoglobin, hematocrit, liver test, lipid test, ketone bodies, 6 uremic toxins (including IS and p-CS), sodium octanoate and decanoate.

SUMMARY:
Current hemodialysis techniques fail to efficiently remove protein-bound uremic toxins (such as p-cresyl sulfate (p-CS) or indoxyl sulfate (IS)) due to their strong binding to serum albumin. The accumulation of these toxins in end-stage renal failure patients on hemodialysis is strongly suspected to contribute to the significant morbidity and mortality observed in this population.

Pre-clinical studies conducted previously showed that medium-chain fatty acids (such as sodium octanoate and decanoate), which are natural ligands of albumin, can effectively displace the binding of uremic toxins on serum albumin and thus promote their elimination during a hemodialysis session.

Medialipide® 20% (Braun) is an emulsion of medium chain triglycerides (MCT) (6 to 12 carbons) used in parenteral nutrition. Medialipide® constitutes a relevant clinical formulation for the administration of octanoate and decanoate because it contains 94% of sodium octanoate and decanoate.

In this study, a proof of concept intervention will be carried out to study the effect on the clearance uremic toxins clearance of the perfusion of Medialipide® emulsion (as a sodium octanoate and decanoate donor) in patients during their hemodialysis session compared to a control situation Sodium chloride (NaCl) 0,9%).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* On haemodialysis at a frequency of 3 sessions of 4 hours per week, for at least 3 months.
* For patients of childbearing age, effective contraception (sexual abstinence, hormonal contraception, intrauterine device or hormone-releasing system, cap, diaphragm or sponge with spermicide, condom) for the entire duration of treatment is required. A blood pregnancy test (beta-human chorionic gonadotropin (HCG)) will be carried out at inclusion.
* Patient affiliated to a social security scheme
* Free, informed and written consent signed by the patient

Exclusion Criteria:

* Residual diuresis > 100 mL per day
* Pregnant or breast-feeding
* Uncontrolled hypertension > 180/115 millimetre of mercury (mmHg)
* Perdialytic hypotension requiring vascular filling > 100 mL during the last 3 sessions
* Patients already on parenteral nutrition
* Patients already on Vitamin K antagonists (VKA) (or prescribed less than one month before inclusion)
* Patients with allergy to heparin or requiring haemodialysis without anticoagulant (recent haemorrhage)
* Criteria relating to products/procedures: Patient with

  * an allergy to egg, soya or peanut proteins or to one of the active ingredients or one of the excipients (glycerol, egg phospholipids for injection, a-tocopherol, sodium oleate (to adjust the pH), water for injection) of Médialipide
  * Severe hyperlipidaemia or severe lipid metabolism disorder characterised by hypertriglyceridaemia > 3 mmol/l
  * Sepsis < 1 month
  * Severe liver failure or cholestasis
  * Known severe coagulopathy
  * Acute thrombo-embolic events
  * Fat embolism
  * Aggravating bleeding diathesis,
  * Uncompensated metabolic acidosis.
  * Unstable circulatory state threatening the vital prognosis (collapse and shock),
  * Unstable metabolic conditions (e.g. severe post-traumatic syndrome, coma of unknown origin),
  * Acute phase of myocardial infarction or stroke,
  * Uncorrected disturbances of fluid and electrolyte balance, such as hypokalaemia and hypotonic dehydration.
  * Decompensated heart failure,
  * Acute pulmonary oedema.
* Subject participating in another interventional study involving a drug with an exclusion period still in progress at inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-22 (Estimated); Study Completion 2027-01-22 (Estimated)

PRIMARY OUTCOMES:
Dialytic clearance of p-CS | until 240 minutes after haemodialysis session
  Dialysis clearance of p-CS (millilitre/minute) is defined as follows:
  Clearance = Qd X (C dialysate/C arterial) with Qd corresponding to the dialysate flow rate, C dialysate the concentration of p-CS in the dialysate, C arterial the concentration of p-CS in the blood sampled at the arterial port of the dialyser.

SECONDARY OUTCOMES:
Reduction fraction (RF) of p-CS | At 240 minutes after haemodialysis session
  Reduction fraction will be measured in percentage Reduction fraction will be compared between the medialipide perfusion situation and the NACL 0,9% perfusion situation.
  RF (%) = (Concentration of p-CS at T0 - Concentration of p-CS at T240)/Concentration of p-CS at T0
Dialytic clearance of Indoxyl sulfate | until 240 minutes after haemodialysis session
  Dialysis clearance of Indoxyl sulfate (millilitre/minute) is defined as follows:
  Clearance = Qd X (C dialysate/C arterial) with Qd corresponding to the dialysate flow rate, C dialysate the concentration of Indoxyl sulfate in the dialysate, C arterial the concentration of Indoxyl sulfate in the blood sampled at the arterial port of the dialyser.
Reduction fraction (RF) of Indoxyl sulfate | At 240 minutes after haemodialysis session
  Reduction fraction will be measured in percentage Reduction fraction will be compared between the medialipide perfusion situation and the NACL 0,9% perfusion situation.
  RF (%) = (Concentration of Indoxyl sulfate at T0 - Concentration of Indoxyl sulfate at T240)/Concentration of Indoxyl sulfate at T0
Dialytic clearance of hippuric acid | until 240 minutes after haemodialysis session
  Dialysis clearance of hippuric acid (millilitre/minute) is defined as follows:
  Clearance = Qd X (C dialysate/C arterial) with Qd corresponding to the dialysate flow rate, C dialysate the concentration of hippuric acid in the dialysate, C arterial the concentration of hippuric acid in the blood sampled at the arterial port of the dialyser.
Reduction fraction (RF) of hippuric acid | At 240 minutes after haemodialysis session
  Reduction fraction will be measured in percentage Reduction fraction will be compared between the medialipide perfusion situation and the NACL 0,9% perfusion situation.
  RF (%) = (Concentration of hippuric acid at T0 - Concentration of hippuric acid at T240)/Concentration of hippuric acid at T0
Dialytic clearance of p-cresyl glucuronide | until 240 minutes after haemodialysis session
  Dialysis clearance of p-cresyl glucuronide (millilitre/minute) is defined as follows:
  Clearance = Qd X (C dialysate/C arterial) with Qd corresponding to the dialysate flow rate, C dialysate the concentration of p-cresyl glucuronide in the dialysate, C arterial the concentration of p-cresyl glucuronide in the blood sampled at the arterial port of the dialyser.
Reduction fraction (RF) of p-cresyl glucuronide | At 240 minutes after haemodialysis session
  Reduction fraction will be measured in percentage Reduction fraction will be compared between the medialipide perfusion situation and the NACL 0,9% perfusion situation.
  RF (%) = (Concentration of p-cresyl glucuronide at T0 - Concentration of p-cresyl glucuronide at T240)/Concentration of p-cresyl glucuronide at T0
Dialytic clearance of indol acetic acid | until 240 minutes after haemodialysis session
  Dialysis clearance of indol acetic acid (millilitre/minute) is defined as follows:
  Clearance = Qd X (C dialysate/C arterial) with Qd corresponding to the dialysate flow rate, C dialysate the concentration of indol acetic acid in the dialysate, C arterial the concentration of indol acetic acid in the blood sampled at the arterial port of the dialyser.
Reduction fraction (RF) of indol acetic acid | At 240 minutes after haemodialysis session
  Reduction fraction will be measured in percentage Reduction fraction will be compared between the medialipide perfusion situation and the NACL 0,9% perfusion situation.
  RF (%) = (Concentration of indol acetic acid at T0 - Concentration of indol acetic acid at T240)/Concentration of indol acetic acid at T0
Dialytic clearance of uric acid | until 240 minutes after haemodialysis session
  Dialysis clearance of indol acetic acid (millilitre/minute) is defined as follows:
  Clearance = Qd X (C dialysate/C arterial) with Qd corresponding to the dialysate flow rate, C dialysate the concentration of uric acid in the dialysate, C arterial the concentration of uric acid in the blood sampled at the arterial port of the dialyser.
Reduction fraction (RF) of uric acid | At 240 minutes after haemodialysis session
  Reduction fraction will be measured in percentage Reduction fraction will be compared between the medialipide perfusion situation and the NACL 0,9% perfusion situation.
  RF (%) = (Concentration of uric acid at T0 - Concentration of uric acid at T240)/Concentration of uric acid at T0
Dialytic clearance of 3-Carboxy-4-methyl-5-propyl-2-furanpropionic acid | until 240 minutes after haemodialysis session
  Dialysis clearance of indol acetic acid (millilitre/minute) is defined as follows:
  Clearance = Qd X (C dialysate/C arterial) with Qd corresponding to the dialysate flow rate, C dialysate the concentration of 3-Carboxy-4-methyl-5-propyl-2-furanpropionic acid in the dialysate, C arterial the concentration of 3-Carboxy-4-methyl-5-propyl-2-furanpropionic acid in the blood sampled at the arterial port of the dialyser.
Reduction fraction (RF) of 3-Carboxy-4-methyl-5-propyl-2-furanpropionic acid | At 240 minutes after haemodialysis session
  Reduction fraction will be measured in percentage Reduction fraction will be compared between the medialipide perfusion situation and the NACL 0,9% perfusion situation.
  RF (%) = (Concentration of 3-Carboxy-4-methyl-5-propyl-2-furanpropionic acid at T0 - Concentration of 3-Carboxy-4-methyl-5-propyl-2-furanpropionic acid at T240)/Concentration of 3-Carboxy-4-methyl-5-propyl-2-furanpropionic acid at T0
Tolerance of medialipide perfusion (%) | until 240 minutes after haemodialysis session
  Percentage of patients with the occurrence of at least one symptom including: nausea, emesis, headaches during the hemodialysis session
Safety of medialipide perfusion | until 7 days after the last haemodialysis session
  % of patients who presented one of the following event : hypertriglyceridemia > 4 gram/liter, alteration of liver test (cytolysis > 2 times the normal value, cholestasis > 2 times the normal value), or hemolysis.
octanoate blood concentration | until 240 minutes after haemodialysis session
decanoate blood concentration | until 240 minutes after haemodialysis session
clearance of octanoate | until 240 minutes after haemodialysis session
  Dialysis clearance of Indoxyl sulfate (millilitre/minute) is defined as follows:
  Clearance = Qd X (C dialysate/C arterial) with Qd corresponding to the dialysate flow rate, C dialysate the concentration of octanoate in the dialysate, C arterial the concentration of octanoate in the blood sampled at the arterial port of the dialyser.
clearance of decanoate | until 240 minutes after haemodialysis session
  Dialysis clearance of Indoxyl sulfate (millilitre/minute) is defined as follows:
  Clearance = Qd X (C dialysate/C arterial) with Qd corresponding to the dialysate flow rate, C dialysate the concentration of decanoate in the dialysate, C arterial the concentration of decanoate in the blood sampled at the arterial port of the dialyser.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Edouard Herriot, Lyon, France